CLINICAL TRIAL: NCT00306306
Title: COOL RCN: Cooling to Prevent Radiocontrast Nephropathy in Patients Undergoing Diagnostic or Interventional Catheterization
Brief Title: COOL RCN: Cooling to Prevent Radiocontrast Nephropathy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radiant Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 50-0212
Record Dates: First submitted 2006-03-21; First posted 2006-03-23 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2007-08

CONDITIONS: Renal Failure; Kidney Failure; Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency

INTERVENTIONS:
Device: Reprieve Endovascular Temperature Therapy System

SUMMARY:
Radiographic contrast agents are administered to all patients undergoing diagnostic or interventional catheterization procedures. Injection of contrast enables visualization of the vasculature with X-ray based fluoroscopy or cineangiographic imaging. Unfortunately, the use of radiographic contrast agents is often associated with severe adverse side effects, including acute kidney failure. Acute kidney failure following exposure to an intravascular contrast agent is also known as Radiocontrast Nephropathy (RCN).

Physiologic factors that may put a patient at higher risk of developing RCN include: pre-existing renal insufficiency, diabetes mellitus, age, cardiovascular disease (particularly congestive heart failure and low ejection fraction), and dehydration or other conditions characterized by depletion of effective circulatory volume. These risk factors are relatively common in patients undergoing catheterization procedures. Treatment of high-risk patients can be modified, by hydration and/or minimizing contrast volume; however despite these efforts, RCN remains a well-recognized complication of coronary catheterization procedures.

Given the frequency and detrimental consequences of RCN, there is a compelling clinical need for safe and effective therapies to reduce the incidence of RCN. One such potential therapy is endovascular cooling to induce mild hypothermia. This study has been designed to evaluate whether endovascular cooling can reduce the incidence of RCN in high-risk patients who are undergoing diagnostic or interventional catheterization procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subject is greater than 18 years of age.
* Subject has a calculated creatinine clearance of 20-50 mL/min (within 10 days prior to enrollment), per the Cockcroft-Gault formula.
* Subject is eligible for coronary angiography (with or without ventriculogram) and/or percutaneous coronary intervention in which it is anticipated that > 50cc of radiographic contrast will be administered.
* Subject agrees to comply with the study procedures, including repeat phlebotomy and clinical follow-up.
* Subject or subject's legal representative is willing to provide written, informed consent to participate in this clinical study.

Exclusion Criteria:

* Subject is currently undergoing renal dialysis.
* Subject is in acute renal failure or has unstable renal function as evidenced by clinical findings or a change in serum creatinine of >= 0.5 mg/dL or >= 25% within 10 days prior to enrollment.
* Subject is undergoing planned renal artery catheterization, or infusion of medications or therapeutic agents directly into the renal arteries.
* Subject is hypotensive [systolic blood pressure (SBP) <100 mmHg].
* Subject has had an acute ST-segment elevation myocardial infarction (MI) within 72 hours prior to enrollment, or is currently having an acute ST-segment elevation MI.
* Subject has decompensated heart failure as defined by the requirement for IV diuretic, inotropic or vasopressor support within the last 7 days.
* Subject requires respiratory support.
* Subject has a known allergy to iodine-based contrast agents that cannot be pre-medicated.
* Subject has received a radiographic contrast agent within 10 days prior to enrollment or a second imaging study is planned within the next 10 days.
* Subject is receiving mannitol or IV diuretics.
* Subject has known renal artery stenosis.
* Subject is currently on a course of chemotherapy.
* Subject has any serious medical condition, which in the opinion of the investigator is likely to interfere with study procedures.
* A plan exists for the addition, discontinuation or dose-adjustment of ACE inhibitors, angiotensin II blockers, trimethoprim, cimetidine, metoclopramide, bromocriptine, levadopa, non-steroidal anti inflammatory drugs (NSAIDs), COX-2 inhibitors, or catechol-O-methyltransferase (COMT) inhibitors (e.g., encapone or tolcapone) at any time during the study.
* Subject has a known hypersensitivity to hypothermia, including a history of Raynaud's Disease.
* Subject has a known hypersensitivity to heparin which cannot be adequately pre-medicated
* Subject has a known history of bleeding diathesis, coagulopathy, sickle cell disease, cryoglobulinemia, or will refuse blood transfusions.
* Subject has a height of < 1.5 m (4 feet 11 inches).
* Subject has an Inferior Vena Cava filter in place.
* Subject is pregnant. (Female subjects of childbearing potential must have a negative serum or urine human chorionic gonadotropin (hCG) pregnancy test prior to enrollment)
* Subject has a known hypersensitivity to buspirone hydrochloride or meperidine and/or has been treated with a monoamine oxidase inhibitor in the past 14 days.
* Subject has a known history of severe hepatic impairment, untreated hypothyroidism, Addison's Disease, or Benign Prostatic Hypertrophy or urethral stricture that in the physician's opinion would be incompatible with meperidine administration.
* Subject has a known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or would be unlikely to comply with study follow-up requirements.
* Subject is currently enrolled in this trial or in another investigational drug or device trial. Note: For the purpose of this protocol, subjects involved in extended follow-up trials for products that were investigational but are currently commercially available are not considered enrolled in an investigational trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-03; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Incidence of RCN
Equivalent safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Gregg Stone, MD, Principal Investigator — Columbia University
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States